CLINICAL TRIAL: NCT05515614
Title: Targeted Nutrition for Moderate to Late Preterm Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 5220169
Record Dates: First submitted 2022-08-19; First posted 2022-08-25 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Premature Birth; Breastmilk Collection; Postnatal Growth Restriction
Keywords: Moderate Preterm; Late Preterm; Postnatal growth; Human milk fortification; Human milk analysis; Targeted nutrition
MeSH Terms: conditions — Premature Birth; Breast Milk Expression

STUDY DESIGN:
Intervention Model Description: Standard nutritional fortification arm (control group): mother's expressed breast milk will be fortified using Enfamil Liquid Human Milk Fortifier (LHMF) as per standard feeding protocol defined by LLUCH NICU Manual.
  In targeted fortification arm (intervention group), mother's expressed breast milk will be fortified with modular components, Amino Acid power, PolyCal and safflower oil, to meet the individual nutritional needs as determined by NICU dieticians.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Mother, physician team, and study statistician will be blinded to randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard Fortification (Active Comparator): Mother's breast milk will be fortified using Enfamil Liquid Human Milk Fortifier (LHMF) as per standard feeding protocol defined by LLUCH NICU.
  Interventions: Dietary Supplement: Enfamil Liquid Human Milk Fortifier
- Targeted Fortification (Experimental): Mother's breast milk will be fortified with modular additives, namely Amino Acid powder, PolyCal, and safflower oil to meet the individual nutritional needs.
  Interventions: Dietary Supplement: Targeted Fortification

INTERVENTIONS:
Dietary Supplement: Targeted Fortification — Mother's breast milk will be fortified in modular fashion based on the level of macronutrients (protein, carbohydrate, and fat) found from analysis using the Miris Human Milk Analyser. For protein supplementation, Amino Acid powder will be utilized as a modular component. For carbohydrate supplementation, PolyCal will be utilized. Mother's breast milk will be fortified in modular fashion. For protein supplementation, Amino Acid powder will be utilized as a modular component. For carbohydrate supplementation, PolyCal will be utilized. For lipid supplementation, safflower oil will be utilized. We will set our goal energy level between 110 - 135 kcal/kg/day, protein level between 3.5 - 4.5 g/kg/day, lipid level between 4.8 - 6.6 g/kg/day, and carbohydrate level between 11.6 - 13.2 g/kg/day. We will regard daily fluid volume to be between 150 to 180 mL/kg/day.
  Arms: Targeted Fortification
Dietary Supplement: Enfamil Liquid Human Milk Fortifier — Mother's breast milk will be fortified using Enfamil Liquid Human Milk Fortifier as per standard feeding protocol defined by LLUCH NICU manual.
  Other Names: LHMF
  Arms: Standard Fortification

SUMMARY:
This study will be comparing the postnatal growth of moderate to late preterm infants in the Neonatal Intensive Care Unit (NICU) born between gestational ages of 30 weeks 0 days to 35 weeks and 6 days who are receiving enteral feeds of mother's own breast milk using the NICU's standard nutritional fortification protocol versus a targeted nutritional fortification protocol.

DETAILED DESCRIPTION:
Infants in the NICU born between gestational ages 30 weeks 0 days and 35 weeks 6 days will be screened to determine if they are receiving unfortified mother's breast milk for enteral nutrition. Informed consent will be obtained from these lactating mothers for themselves and their infants to participate in the study. Once enrolled in the study, the mother and infant dyad will be randomized using an electronic tool for block randomization into standard fortification arm (control group) or targeted fortification arm (intervention group). Maximum of 100 infants will be assigned to each arm to ensure statistical significance. The physician team, study statisticians, and the mothers will be blinded in their group assignment.

Mothers will be provided with one-on-one teaching (with verbal and written instructions) by the NICU certified lactation consultants or by an authorized, trained study personnel on how to pool their pumped breast milk for 24 hours, referenced as "breast milk pooling." They will also be shown how to prepare a 10 mL sample of the pooled breast milk for analysis. Pooled breast milk will be analyzed for macronutrient content (protein, carbohydrate, fat, and calories) using Miris Human Milk Analyzer before fortification once a week for both arms of the study. All infants in both groups will follow the enteral feeding advancement schedule until the infant is ready for nutritional fortification.

In the standard fortification arm (control group), mother's breast milk will be fortified using Enfamil Liquid Human Milk Fortifier (LHMF) as per standard feeding protocol defined by Loma Linda University Children's Hospital Neonatal Intensive Care Unit. The feeding protocol, specific to birth weight, is available online in the LLUCH NICU Manual.

In the targeted fortification arm (intervention group), mother's breast milk will be fortified in modular fashion. For protein supplementation, Amino Acid powder will be utilized as a modular component. For carbohydrate supplementation, PolyCal will be utilized. For lipid supplementation, safflower oil will be utilized. Fortification goals for this group will follow the macronutrient intake recommendations for preterm infants published by the European Society of Paediatric Gastroenterology, Hepatology and Nutrition (ESPGHAN) Committee on Nutrition in 2009. The goal energy level will be between 110 - 135 kcal/kg/day, goal protein level between 3.5 - 4.5 g/kg/day, goal lipid level between 4.8 - 6.6 g/kg/day, and goal carbohydrate level between 11.6 - 13.2 g/kg/day. The goal total daily fluid volume will be between 150 to 180 mL/kg/day.

NICU Registered Dietitians will be provided with the macronutrient contents of pooled breast milk from mothers of babies in the intervention group. Using the aforementioned values from ESPGHAN guideline for each macronutrient, they will provide recommendations on specific amounts of modular supplementation to be added to the pooled breast milk. Based on these recommendations, all un-pooled expressed breast milk of mothers in the intervention group will be fortified in a customized manner by the milk technicians in the NICU milk room and given to infants in the intervention group. NICU Registered Dieticians will not be provided with analysis results showing macronutrient levels of the pooled milk or standard fortified milk in the control group as the current standard of care at LLUCH NICU does not include macronutrient analysis of pooled breast milk for babies born >30 weeks gestation.

Infants enrolled in both arms will have their anthropometric measurements taken once a week from birth to NICU discharge. Anthropometric measurements will include weight, height, and head circumference. The Z-scores of weight, height, and head circumference will be recorded and analyzed for any statistical differences.

ELIGIBILITY:
Inclusion Criteria:

* Singleton preterm infants
* Between 30 weeks 0 days and 35 weeks and 6 days
* Receiving any amount of mother's breast milk as a form of enteral nutrition
* Mother is ≥ 18 y/o

Exclusion Criteria:

* Not receiving any breast milk
* Congenital anomalies or surgical conditions that interfere with enteral feeding

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2022-08-17 (Actual); Primary Completion 2023-05-11 (Actual); Study Completion 2023-05-11 (Actual)

PRIMARY OUTCOMES:
Postnatal growth in weight | From date of birth to date of NICU discharge or when breast milk is no longer available, whichever comes first, assessed up to 24 months
  Weight in kilograms
Postnatal growth in length | From date of birth to date of NICU discharge or when breast milk is no longer available, whichever comes first, assessed up to 24 months
  Length in centimeters
Postnatal growth in head circumference | From date of birth to date of NICU discharge or when breast milk is no longer available, whichever comes first, assessed up to 24 months
  Head circumference in centimeters
Protein level in mother's expressed breastmilk | From date of first breast milk analysis to date of NICU discharge or when breast milk is no longer available, whichever comes first, assessed up to 24 months
  Weekly analysis of pooled mother's expressed breast milk to assess for protein level, measured in grams per 100 milliliters
Calories in mother's expressed breastmilk | From date of first breast milk analysis to date of NICU discharge or when breast milk is no longer available, whichever comes first, assessed up to 24 months
  Weekly analysis of pooled mother's expressed breast milk to assess for amount of calories, measured in kilocalories per 100 milliliters
Fat content in mother's expressed breastmilk | From date of first breast milk analysis to date of NICU discharge or when breast milk is no longer available, whichever comes first, assessed up to 24 months
  Weekly analysis of pooled mother's expressed breast milk to assess for fat content, measured in grams per 100 milliliters
Carbohydrate level in mother's expressed breastmilk | From date of first breast milk analysis to date of NICU discharge or when breast milk is no longer available, whichever comes first, assessed up to 24 months
  Weekly analysis of pooled mother's expressed breast milk to assess for carbohydrate level, measured in grams per 100 milliliters

CONTACTS AND LOCATIONS:
Overall Officials: Raylene Phillips, MD, Principal Investigator — Loma Linda University
Locations (1):
- Loma Linda University, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shapiro-Mendoza CK, Tomashek KM, Kotelchuck M, Barfield W, Nannini A, Weiss J, Declercq E. Effect of late-preterm birth and maternal medical conditions on newborn morbidity risk. Pediatrics. 2008 Feb;121(2):e223-32. doi: 10.1542/peds.2006-3629. PMID 18245397
- [Background] Radtke JV. The paradox of breastfeeding-associated morbidity among late preterm infants. J Obstet Gynecol Neonatal Nurs. 2011 Jan-Feb;40(1):9-24. doi: 10.1111/j.1552-6909.2010.01211.x. PMID 21244492
- [Background] Al-Theyab NA, Donovan TJ, Eiby YA, Colditz PB, Lingwood BE. Fat trajectory after birth in very preterm infants mimics healthy term infants. Pediatr Obes. 2019 Mar;14(3):e12472. doi: 10.1111/ijpo.12472. Epub 2018 Sep 26. PMID 30257276
- [Background] Chmielewska A, Farooqi A, Domellof M, Ohlund I. Lean Tissue Deficit in Preterm Infants Persists up to 4 Months of Age: Results from a Swedish Longitudinal Study. Neonatology. 2020;117(1):80-87. doi: 10.1159/000503292. Epub 2019 Dec 10. PMID 31822002
- [Background] Rochow N, Fusch G, Ali A, Bhatia A, So HY, Iskander R, Chessell L, El Helou S, Fusch C. Individualized target fortification of breast milk with protein, carbohydrates, and fat for preterm infants: A double-blind randomized controlled trial. Clin Nutr. 2021 Jan;40(1):54-63. doi: 10.1016/j.clnu.2020.04.031. Epub 2020 May 6. PMID 32446787
- [Background] Chou FS, Yeh HW. Sex differences in postnatal weight gain trajectories of extremely preterm newborns. J Perinatol. 2021 Aug;41(8):1835-1844. doi: 10.1038/s41372-021-01099-2. Epub 2021 May 25. PMID 34035451
- [Background] Agostoni C, Buonocore G, Carnielli VP, De Curtis M, Darmaun D, Decsi T, Domellof M, Embleton ND, Fusch C, Genzel-Boroviczeny O, Goulet O, Kalhan SC, Kolacek S, Koletzko B, Lapillonne A, Mihatsch W, Moreno L, Neu J, Poindexter B, Puntis J, Putet G, Rigo J, Riskin A, Salle B, Sauer P, Shamir R, Szajewska H, Thureen P, Turck D, van Goudoever JB, Ziegler EE; ESPGHAN Committee on Nutrition. Enteral nutrient supply for preterm infants: commentary from the European Society of Paediatric Gastroenterology, Hepatology and Nutrition Committee on Nutrition. J Pediatr Gastroenterol Nutr. 2010 Jan;50(1):85-91. doi: 10.1097/MPG.0b013e3181adaee0. PMID 19881390
- See also: CDC Wonder Natality, 2016-2020 — https://wonder.cdc.gov/natality.html